CLINICAL TRIAL: NCT06391515
Title: Subacute Thyroiditis in the SARS-CoV-2 Era: a Multicentre Prospective Study
Brief Title: Subacute Thyroiditis in the SARS-CoV-2 Era
Acronym: SAT-COVID-19
Status: Completed | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Giulia Brigante, MD, PhD, University of Modena and Reggio Emilia
Other Study IDs: 1104/2020
Record Dates: First submitted 2024-04-29; First posted 2024-04-30 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Subacute Thyroiditis; SARS CoV 2 Infection; Thyrotoxicosis
MeSH Terms: conditions — Thyroiditis, Subacute; COVID-19; Thyrotoxicosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid +: At baseline, a blood sample was collected and centrifuged for serological analysis. Then, sera were stored at -20°C until the end of the enrolment phase when all samples were centralized at the coordinating center for SARS-CoV-2 IgG measurements. IgG against the spike protein (anti-S IgG) and against nucleocapside (anti-N IgG) were tested. Anti-N IgG increase only after natural infection since the nucleocapsid protein is not contained in the vaccines, while anti-S IgG increase is induced either by vaccination or infection 21. Thus, we subdivided patients according to their serological status: i) group Covid+ included those patients who had both positive anti-S and anti-N IgG demonstrating a contact with SARS-CoV-2 before the diagnosis of SAT; ii) group Covid- consisted of patients with only anti-S IgG positivity (due to vaccine) or negative anti-N/anti-S IgG.
  Interventions: Diagnostic Test: Blood sample, CRF, thyroid ultrasound
- Covid -: At baseline, a blood sample was collected and centrifuged for serological analysis. Then, sera were stored at -20°C until the end of the enrolment phase when all samples were centralized at the coordinating center for SARS-CoV-2 IgG measurements. IgG against the spike protein (anti-S IgG) and against nucleocapside (anti-N IgG) were tested. Anti-N IgG increase only after natural infection since the nucleocapsid protein is not contained in the vaccines, while anti-S IgG increase is induced either by vaccination or infection 21. Thus, we subdivided patients according to their serological status: i) group Covid+ included those patients who had both positive anti-S and anti-N IgG demonstrating a contact with SARS-CoV-2 before the diagnosis of SAT; ii) group Covid- consisted of patients with only anti-S IgG positivity (due to vaccine) or negative anti-N/anti-S IgG.
  Interventions: Diagnostic Test: Blood sample, CRF, thyroid ultrasound

INTERVENTIONS:
Diagnostic Test: Blood sample, CRF, thyroid ultrasound — Five visits were planned: at diagnosis (V0) and after 1, 3, 6 and 12 months (V1, V2, V3 and V4, respectively). At each visit, subjects were evaluated with anamnesis, physical examination, thyroid US and blood tests.

SUMMARY:
Many cases of subacute thyroiditis (SAT) have been described related to SARS-CoV-2 infection, but no prospective data about follow-up is known. This prospective, longitudinal, 3-year, multicentre study is aimed at exploring clinical peculiarities and outcome of SAT in relation to SARS-CoV-2 infection, ascertained with antibody dosage.

All patients receiving SAT diagnosis from November 2020 to May 2022 were enrolled. Multicentre study. Data about anamnesis, physical examination, blood tests (TSH, freeT4, freeT3, thyroglobulin, anti-thyroid antibodies, C-reactive protein, erythrocyte sedimentation rate, complete blood count), and thyroid ultrasound were collected. At baseline, the presence of IgG against the SARS-CoV-2 spike protein or nucleocapside was investigated. Patients were evaluated after 1, 3, 6, 12 months.

DETAILED DESCRIPTION:
A multicentre, longitudinal, prospective study was conducted, enrolling all patients diagnosed with SAT at the participating centres between November 2020 and May 2022. The following Italian centres participated: Endocrinology Unit of Azienda Ospedaliero-Universitaria of Modena (Coordinating center); Endocrinology Unit of IRCCS Ca' Granda Ospedale Maggiore Policlinico of Milano; Endocrinology and Diabetes Prevention and Care Unit of the IRCCS Azienda Ospedaliero-Universitaria Policlinico of Bologna. These Units were involved through a call launched by the coordinating center to the young Italian members of the Club EnGioI (Endocrinologia Giovane in Italia) of the Italian Society of Endocrinology (SIE).

Five visits were planned: at diagnosis (V0) and after 1, 3, 6 and 12 months (V1, V2, V3 and V4, respectively). At each visit, subjects were evaluated with anamnesis, physical examination, thyroid ultrasound and blood tests. Patients were treated according to the clinical presentation and to the current guidelines. Nonsteroidal anti-inflammatory drugs (NSAIDs) were preferred in patients with mild symptoms and mild laboratory findings; steroid therapy was preferred in those with severe symptoms and/or those who did not respond to NSAIDs within 1 to 2 weeks. Beta-blockers were prescribed as symptomatic treatment in case of tachycardia. During the follow-up phase, the therapeutic approach and any change of it were recorded.

Finally, the treatment responsiveness and outcomes of transient hypothyroidism, permanent hypothyroidism, or recurrence during the follow-up period were all documented.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of subacute thyroiditis
* age ≥ 18 years
* willingness to sign an informed consent

Exclusion Criteria:

* ongoing pregnancy
* alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with clinical diagnosis of SAT were enrolled. Diagnosis was made by experienced endocrinologists according to guidelines 2: thyroid tenderness and anterior neck pain, often radiating to ears, jaw, or throat, spreading from one side to the other, low-grade fever, pharyngitis symptoms, fatigue, thyroid slightly enlarged, firm and painful to palpation, ESR or CRP elevation.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
quantification of neck pain at diagnosis | at diagnosis
  evaluation in a scale from 0 to 10 (10 means maximum pain)
description of neck pain at diagnosis | at diagnosis
  localization at right or left side, migrating, radiating to the ears
duration of neck pain at diagnosis | at diagnosis
  duration in days

SECONDARY OUTCOMES:
quantification of neck pain at follow-up | 1, 3, 6 and 12 months after diagnosis
  evaluation in a scale from 0 to 10 (10 means maximum pain)
description of neck pain at follow-up | 1, 3, 6 and 12 months after diagnosis
  localization at right or left side, migrating, radiating to the earsmaximum pain)
duration of neck pain at follow-up | 1, 3, 6 and 12 months after diagnosis
  duration in days
thyroid inhomogeneity at ultrasound | at diagnosis and after1, 3, 6 and 12 months
  US examination performed by endocrinologists with at least 5 years of experience in US neck examination with a linear probe. SAT-related findings such as inhomogeneity will be evaluated (present or absent)
thyroid function at diagnosis and follow-up | at diagnosis and after1, 3, 6 and 12 months
  thyroid stimulating hormone (TSH), free thyroxine (fT4), free triiodothyronine (fT3), thyroglobulin (Tg), thyroglobulin antibodies (TgAb), anti-thyroid peroxidase antibodies (TPOAb), thyrotropin receptor antibodies (TRAb)
thyroid stimulating hormone (TSH) serum levels at diagnosis and follow-up | at diagnosis and after1, 3, 6 and 12 months
  thyroid stimulating hormone (TSH) serum levels
free thyroxine (fT4) at diagnosis and follow-up | at diagnosis and after1, 3, 6 and 12 months
  free thyroxine (fT4) serum levels
free triiodothyronine (fT3) at diagnosis and follow-up | at diagnosis and after1, 3, 6 and 12 months
  free triiodothyronine (fT3) serum levels
thyroglobulin (Tg) at diagnosis and follow-up | at diagnosis and after1, 3, 6 and 12 months
  thyroglobulin (Tg) serum levels
thyroglobulin antibodies (TgAb) at diagnosis and follow-up | at diagnosis and after1, 3, 6 and 12 months
  thyroglobulin antibodies (TgAb) serum levels
anti-thyroid peroxidase antibodies (TPOAb) at diagnosis and follow-up | at diagnosis and after1, 3, 6 and 12 months
  anti-thyroid peroxidase antibodies (TPOAb) serum levels
thyrotropin receptor antibodies (TRAb) at diagnosis and follow-up | at diagnosis and after1, 3, 6 and 12 months
  thyrotropin receptor antibodies (TRAb) serum levels

CONTACTS AND LOCATIONS:
Locations (1):
- University of Modena and Reggio Emilia, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided